CLINICAL TRIAL: NCT03558373
Title: The Adherence of Immunosuppressive Therapy Including Tacrolimus Once Daily in a Cohort of Kidney Transplant Recipients: an Italian Prospective Observational Study
Brief Title: The Adherence of Immunosuppressive Therapy Including Tacrolimus Once-daily in Italian Kidney Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: DFIDM-1701
Record Dates: First submitted 2018-05-28; First posted 2018-06-15 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Kidney Transplant
Keywords: adherence; tacrolimus; once-daily
MeSH Terms: interventions — Immunosuppressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Immunosuppressive — Immunosuppressive therapies

SUMMARY:
Non-adherence is widespread in the transplant community. Addressing issues associated with non-adherence remains a key challenge in transplantation, in part due to the difficulty in assessing its prevalence, as there is currently no 'gold standard' for use in routine clinical practice.

The purpose of this study is to evaluate the non-adherence to immunosuppressive therapy, including tacrolimus once-daily, among Italian kidney transplant recipients receiving. Along with non-adherence evaluation, possible factors related to NA will be investigated (patient-related, condition/disease-related, therapy/treatment-related, etc.).

ELIGIBILITY:
Inclusion criteria:

1. Adult (≥ 18 years) recipients of a deceased- or living-donor kidney transplant since maximum 12 months.
2. Recipients with a functioning graft
3. Patients receiving tacrolimus once-daily as part of their IS therapy since minimum 2 months.
4. Patients who have signed informed consent form and privacy form.
5. Patients capable of discernment and able to read and write in Italian language.

Exclusion criteria:

1. Patients received or planned to receive, a non-renal solid organ transplant, a simultaneous pancreas-kidney transplant, or a bone narrow transplant.
2. Patients who already received a kidney transplant (re-transplant).
3. Patients enrolled or planned to be enrolled in any clinical study.
4. Patients suffering from conditions and illnesses that might interfere with the study purpose, according to the investigator's evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Non aderence | 6 months
  Proportion of non-adherent patients to immunosuppressive therapy as measured by the Basel Assessment of Adherence with Immunosuppressives Scale (BAASIS©-interview). The BAASIS© consists of four items (with a 6-point scale for responses ranging from never (0) to every day (5)) measuring patients' taking, skipping (or drug holidays), timing (>2 hrs from prescribed time) and dose reduction of drugs. An affirmative answer to any of the first 4 questions results in assignment to the non-adherent group.

SECONDARY OUTCOMES:
BMQ score | Baseline and 6 months
  Describe the patient's belief about immunosuppresive medicines, as measured by the Belief about Medicines Questionnaire (BMQ). It is an 18-item measure comprising of two subscales (general harm and general overuse), and two subscales (specific necessity and specific concerns). Higher scores in the General-Harm and General-Overuse sub-scales represent an overall negative perception of medication. High scores in the Specific-Concerns sub-scale means that adverse reactions are potentially harmful and high scores in the Specific-Necessity sub-scale are indicative of the patient's need to adhere to medication to maintain health.
ACCEPT score | Baseline and 6 months
  Describe the patient's acceptance toward immunosuppressive treatment, as measured by the ACCEPT questionnaire. It is a 32-items self-administered questionnaire and covers patient's opinion on: convenience of the medication, length of treatment, constraints due to medication, side effects and a general opinion on the medication. The score ranges from 0 (no acceptance) to 100 (maximum treatment acceptance).
BAASIS evaluation | Baseline
  Perform the BAASIS assessement.The BAASIS consists of four items (with a 6-point scale for responses ranging from never (0) to every day (5)) measuring patients' taking, skipping (or drug holidays), timing (>2 hrs from prescribed time) and dose reduction of drugs. An affirmative answer to any of the first 4 questions results in assignment to the non-adherent group.
Patients characteristics | Baseline
  Describe patients characteristics (such as socio-demographics, lifestyle information, relevant comorbidities, concomitant medications, clinical characteristics information like e.g. primary kidney disease diagnosis, waiting time before graft, transplant characteristic e.g. type of donor, etc.
Clinical informations as for clinical practice | Baseline and 6 months
  Collect clinical information (e.g. routine tacrolimus trough levels, eGFR if available)
Immunosuppressive treatments | Baseline and 6 months
  Immunosuppressive treatments description and changes
Rejections | Baseline and 6 months
  Occurrence of rejection episodes
Graft failure | Baseline and 6 months
  Occurrence of graf failure
Adverse events | Baseline and 6 months
  Number of adverse events
Infections | Baseline and 6 months
  Occurrence of infections
Healthcare cost | 6 months
  Assess the healthcare cost (ER admission, hospitalizations)

CONTACTS AND LOCATIONS:
Locations (12):
- Italy (12):
  - A.O.U. Consorziale Policlinico, Bari
  - A.O.U. Policlinico S.Orsola Malpighi, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - A.O.U. Maggiore della Carità, Novara
  - Azienda Ospedaliera di Padova, Padua
  - ARNAS Ospedale Civico, Palermo
  - A.O.U. Pisana P.O. Cisanello, Pisa
  - Ospedale Cisanello, Pisa
  - Fondazione Policlinico Univ. Gemelli, Roma
  - A.O.U. Città della Salute e della Scienza, Torino
  - A.O. Ospedale Circolo e Fondazione Macchi, Varese
  - A.O.U.I. Ospedale Borgo Trento, Verona

IPD SHARING:
Plan to Share IPD: No